CLINICAL TRIAL: NCT01600482
Title: Clinical Investigation Plan (CIP) for Safety and Efficacy Study of Arterial Closure Device (CELT ACD). Clinical Investigation Plan No.: CIP-TS-003
Brief Title: Clinical Investigation for Safety and Efficacy Study of CELT ACD (Arterial ClosureDevice)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vasorum Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP-TS-003
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Disease; Coronary Artery Disease
Keywords: Hemostasis.; Percutaneous coronary interventions.; Closure Device
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CELT ACD device (Experimental): The CELT ACD device is a vascular closure device.
  Interventions: Device: CELT ACD
- Manual Compression (No Intervention): Manual Compression

INTERVENTIONS:
Device: CELT ACD — The CELT ACD will be used to achieve hemostasis of the common femoral artery in patients on anticoagulation who are undergoing a percutaneous intervention procedure using a 6F procedural sheath.
  Arms: CELT ACD device

SUMMARY:
The objective of the CELT ACD® Vascular Closure Device study is to evaluate the safety and effectiveness of the CELT ACD® device to achieve hemostasis of the common femoral artery access site in patients on anticoagulation who are undergoing a percutaneous intervention (PCI) procedure using a 6F sheath.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age.
2. Each patient, or his or her guardian or legal representative, is willing to give informed consent.
3. Clinically indicated for an intra-arterial procedure involving access through the common femoral artery and conducted through an access sheath size of between 6F and 7F inclusive.

Exclusion Criteria:

1. Patients with known allergy to any of the materials used in the device.
2. Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than one year.
3. Evidence of systemic bacterial or cutaneous infection, including groin infection.
4. Patients suffering with definitive or potential coagulopathy or platelet count <100,000./µl
5. Use of systemic thrombolytic agents within 24 hours prior to or during the catheterization procedure which cause the concentration of fibrinogen to be < 100 mg/dl or if post-thrombolytic fibrinogen (in case of thrombolysis within 24 hours or intra-procedural) cannot be measured.
6. Patients in whom an introducer sheath smaller than 6F or greater than 7F have been used.
7. Currently participating in another investigational device or drug study.
8. Patients with severe claudication, iliac or femoral artery diameter stenosis greater than 50%, or previous bypass surgery or stent placement in the vicinity of the access site.
9. If puncture site is via a vascular graft.
10. If a palpable haematoma is observed during the procedure.
11. Patients in whom there is any indication that puncture has been made in the profunda femorals artery or superficial femoral artery, or adjacent to the bifurcation.
12. Patients with a common femoral artery lumen diameter of less than 5 mm.
13. Patients that have any amputation from an access site limb.
14. Patients that have undergone a percutaneous procedure using a vascular closure device for hemostasis within the previous 30 days or using manual/mechanical pressure for hemostasis within the prior 30 days in the same leg.
15. Patients with a systolic blood pressure reading below 90 mmHg.
16. Patients with an active haematoma, arteriovenous fistula, or pseudoaneurysm.
17. Patients with a very superficial artery where the depth from skin to the artery surface at the access site is less than 4 mm.
18. Morbidly obese patients (Body Mass Index >35kg/m2).
19. Patients with a stent less than or equal to 1 cm of the puncture site that would interfere with placement of the device implant.
20. Patient is know or suspected to be pregnant, or is lactating.
21. Patients in whom there has been an antegrade puncture.
22. Patients in whom there has been difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial wall puncture.
23. Patients who have undergone prior or recent use of an intra-aortic balloon pump through the arterial access site.
24. Patients with uncontrolled hypertension (BP greater than or equal to 180/110mmHg) at time of vascular closure
25. Patients with acute ST-elevation myocardial infarction less than or equal to 48hours before catheterization procedure.
26. Patients with cardiogenic shock (hemodynamic instability requiring intravenous medication or mechanical support) experienced during or immediately post-catheterization.
27. Patients who are unable to ambulate at baseline.
28. Patients known to require an extended hospitalization (e.g. patient is undergoing cardiac surgery).
29. Patient has already participated in the trial.
30. Patient is unavailable for follow up.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - New York Presbyterian Hospital, New York, New York
- Germany (2):
  - Städtische Kliniken Neuss - Lukaskrankenhaus - GmbH, Preußenstr. 84,41464 Neuss, Neuss
  - Charite Campus Mitte, Berlin
- Galway University Hosptial, Galway, Ireland, Ireland

REFERENCES:
- [Derived] Wong SC, Laule M, Turi Z, Sanad W, Crowley J, Degen H, Bennett K, Coleman JE, Bergman G. A multicenter randomized trial comparing the effectiveness and safety of a novel vascular closure device to manual compression in anticoagulated patients undergoing percutaneous transfemoral procedures: The CELT ACD trial. Catheter Cardiovasc Interv. 2017 Nov 1;90(5):756-765. doi: 10.1002/ccd.26991. Epub 2017 Mar 15. PMID 28296003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per agreement with FDA, following the 207 patient 6F Celt ACD study, an additional 34 patients were recruited across 3 clinical investigation sites whereby a 7F Celt ACD device was used to close an arterial puncture made with a 7F sheath in fully anti-coagulated patients. 7F device approval is pending with FDA.
Groups:
- CELT ACD Device: The CELT ACD device is a vascular closure device.
  CELT ACD: The CELT ACD will be used to achieve hemostasis of the common femoral artery in patients on anticoagulation who are undergoing a percutaneous coronary intervention procedure using either a 6F or a 7F procedural sheath.
Period: Overall Study
Arm/Group | CELT ACD Device | Manual Compression
Started | 148 | 59 (Last 26 patients allocated to CELT ACD)
Completed | 148 (Last 26 patients allocated to CELT ACD) | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CELT ACD Device | Manual Compression | Total
Number analyzed (Participants) | 148 | 59 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.75 (10.8) | 67.44 (11.7) | 66.95 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 12 | 48
  Male | 112 | 47 | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 20 | 57
  Ireland | 69 | 21 | 90
  Germany | 42 | 18 | 60
Weight [Mean (Standard Deviation); unit: Kgs] | 85.38 (16.22) | 82.78 (40.83) | 84.65 (15.80)
Height [Mean (Standard Deviation); unit: cm] | 172.90 (9.56) | 171.70 (7.82) | 172.50 (9.12)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.75 (4.47) | 28.18 (4.41) | 27.87 (4.45)
Right Femoral Artery Site [Count of Participants; unit: Participants] | 142 | 57 | 199

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint Will be the Combined Rate of Major Complications With in 30 +/- 7 Days Following the Percutaneous Coronary Intervention (PCI) Procedure.
Description: rate of major complications with in 30 +/- 7 days following the PCI procedure.
Time Frame: With in the first 30 days +/- 7 days following the procedure
Measure: Number; unit: major complications
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 148 | 59
major complications | 1 | 2

2. Primary Outcome: The Primary Effectiveness Endpoint Will be Time to Hemostasis (TTH)
Description: Time to hemostasis
Time Frame: With in the first 30 days +/- 7 days following the procedure
Population: 7 subjects in manual compression group where TTH was not recorded.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 148 | 52
minutes | 0.99 (4.15) | 17.54 (54.55)

3. Secondary Outcome: The Secondary Safety Endpoint Will be the Combined Rate of Minor Complications With in 30 +/- 7 Days Following Procedure.
Description: combined rate of minor complications with in 30 +/- 7 days following procedure.
Time Frame: With in the first 30 days +/- 7 days following the procedure
Measure: Number; unit: minor complications
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 148 | 59
minor complications | 7 | 5

4. Secondary Outcome: Time to Ambulation
Description: Time to Ambulation (TTA) is defined as the time elapsed between sheath removal and time when the patient stands and walk 6m (20ft) without re-bleeding.
Time Frame: With in the first 30 days +/- 7 days following the procedure
Population: 62 patients did not have TTA recorded.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 101 | 44
minutes | 360.0 (418.4) | 406.4 (216.2)

5. Secondary Outcome: Time to Discharge-ability
Description: Time to discharge-ability
Time Frame: 30 days +/- 7 days
Population: 107 did not have time to dischargeability data collected.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 71 | 29
Minutes | 662.51 (511.70) | 511.76 (350.2)

6. Secondary Outcome: Procedure Success
Description: Procedure Success 30 days +/- 7 days
Time Frame: 30 days +/- 7 days
Population: 7 patients were excluded in Manual Compression group as there was no TTH data recorded.
Measure: Number; unit: Number of patients
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 148 | 52
Number of patients | 147 | 51

7. Secondary Outcome: Device Success
Description: Device Success (DS) is defined as the successful deployment of the Celt ACD device with the attainment of haemostasis and only assessed in the Celt ACD arm of the study.
Time Frame: 30 days +/- 7 days
Population: 7 patients in the MP group did not have TTH recorded.
Measure: Number; unit: Number of patients
Arm/Group | CELT ACD Device | Manual Compression
Number analyzed (Participants) | 148 | 0
Number of patients | 147 |

ADVERSE EVENTS:
Time Frame: 30 days +/- 7 days
Arm/Group | CELT ACD Device | Manual Compression
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/148 | 2/59
Other Adverse Events (participants affected / at risk) | 0/148 | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CELT ACD Device (N=148) | Manual Compression (N=59)
Device migration (Surgical and medical procedures) | 1 (1) | 0 (0) — Device migration from femoral artery access point
Syncope (Surgical and medical procedures) | 0 (0) | 1 (1) — Syncope during the follow up period
Brain Stem Ischemia (Vascular disorders) | 0 (0) | 1 (1) — Brain stem ischemia unrelated to procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No